CLINICAL TRIAL: NCT01023854
Title: Consideration of the Merits of Continuous Paravertebral Block in the Management of Renal and/or Adrenal Surgery by Laparotomy in Adults
Brief Title: Merits of Continuous Paravertebral Block in the Management of Renal/Adrenal Surgery by Laparotomy
Acronym: BPV
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No more potentiel patients for study
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BPV; RB 09.011 (Registry Identifier: AFSSAPS A90622-20)
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Indication for Renal and/or Adrenal Surgery
Keywords: Paravertebral block; loco regional anesthesia; renal surgery; PCA morphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Continuous Paravertebral block (Experimental): Continuous Paravertebral block
  Interventions: Procedure: Continuous Paravertebral block
- Placebo (Placebo Comparator): Placebo
  Interventions: Procedure: Continuous Paravertebral block

INTERVENTIONS:
Procedure: Continuous Paravertebral block — The paravertébral block is a peripheral block which gets an one-sided continuous analgesia by infiltration of the spinal nerves which appear from the intervertebral foramen.
  Its realization consists of a draining in 2-3 cm of the thorny apophyses ( T6-T8). During the perception of the osseous contact (cross-functional process of the vertebra), the needle is redirected in cephalic direction until a loss of resistance corresponding to the passage of the upper costo-cross-functional ligament that is in the entrance to the paravertébral space. A catheter is then inserted into the paravertébral space.

SUMMARY:
The paravertebral block is an alternative in the analgesia epidural the major interest of which lives in the catheterisation of the paravertébral space allowing to assure/insure an one-sided continuous analgesia.

The main objective of the study is to bring to light the superiority of the continuous paravertébral block, as a supplement to analgesia, in the care of the renal and\or adrenal surgery by laparotomy at the adult in terms of consumption of morphine, with regard to the classic analgesia classic.

The main assessment criterion is the consumption of morphine within first 24 postoperative hours at the patients benefiting from a paravertébral continuous block besides the classic systematic analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patient scheduled for renal and/or adrenal surgery
* American Society of Anesthesiologists score ASA I, II, III
* Written informed consent given by the patient

Exclusion Criteria:

* Contraindication in the loco-regional anesthesia in the products of local anesthetic
* Surgery as a matter of urgency
* Pregnancy
* Congestive Cardiac insufficiency
* Severe hepatic Incapacity
* Disturbs of the coagulation
* Age < 18 years
* ASA IV
* Patient already participating in a study or deadline 3-month-old subordinate since the end of a previous study
* Under guardianship Patient
* Psychiatric pathology or limitation of the intellectual abilities making difficult the understanding of the subjective questions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-10; Primary Completion 2012-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
morphine consumption during the first 24 hours | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: François LION, Doctor, Principal Investigator — Brest, Hospital University
Locations (1):
- Cavale Blanche Hospital, Brest, France